CLINICAL TRIAL: NCT02565576
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Preliminarily Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of CFZ533 in Patients With Moderate to Severe Myasthenia Gravis
Brief Title: Safety,Tolerability,Pharmacokinetics and Efficacy of CFZ533 in Moderate to Severe Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCFZ533X2204
Record Dates: First submitted 2015-06-23; First posted 2015-10-01 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-07

CONDITIONS: Myasthenia Gravis, Generalized
Keywords: CFZ533, Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — iscalimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CFZ533 (Active Comparator): CFZ533
  Interventions: Drug: Placebo; Drug: CFZ533
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
Drug: CFZ533
  Arms: CFZ533

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, pharmacokinetics/pharmacodynamics and efficacy of CFZ533 as an add-on therapy to standard of care in patients with moderate to severe myasthenia gravis (MG).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MG class IIa to IVa inclusive (Myasthenia Gravis Foundation of America Clinical Classification).
2. Quantitative Myasthenia Gravis (QMG) score of 10 or greater. If the QMG score is < 15 no more than 4 points may be derived from items 1 or 2 (ocular motility disturbance and ptosis).
3. Documented history of acetylcholine receptor (AChR) or Muscle Specific Kinase (MuSK) antibody positive.
4. Only one immunosuppressant or immunomodulatory drug at a stable dose is allowed during the study (i) azathioprine and mycophenolate mofetil must be stable for at least 4 months prior to randomization (ii) cyclosporine must be stable for at least 3 months prior to randomization.
5. If the patient is on oral corticosteroids, methotrexate or tacrolimus at screening, the dose must be stable for at least 1 month prior to randomization.
6. If the patient is on cholinesterase inhibitors at screening, the dose must be stable for at least 2 weeks prior to randomization.
7. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, may be included in the study if they are using highly effective methods of contraception during the study and for 12 weeks after study treatment.

Exclusion Criteria:

1. MGFA grade I, IVb, or V disease.
2. Documented presence of unresected thymoma.
3. Patients having undergone thymectomy or thymo thymectomy (resection of thymoma) within 6 months of screening.
4. Patients having received any of the following treatments prior to randomization:

   1. IVIg or plasma exchange within 8 weeks;
   2. oral or IV cyclosphosphamide treatment within 3 months;
   3. IV corticosteroid bolus (dose higher than 1 mg/kg) within 3 months;
   4. belimumab within 6 months. For patients who received belimumab earlier, B cell count should be within normal range;
   5. rituximab within 12 months. For patients who received rituximab earlier, B cell count should be within normal range;
   6. any other biologic or an investigational drug within 1 month or five times thehalf-life, whichever is longer.
   7. Live vaccines within 4 weeks of study drug infusion.
5. Patients who are at significant risk for TE as judged by the investigator or have any one of the following:

   1. History of either thrombosis or 3 or more spontaneous abortions with or without the presence of anti-cardiolipin autoantibodies;
   2. Presence of prolonged partial thromboplastin time (PTT).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Canada (2):
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Denmark (2):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Halle/S
  - Novartis Investigative Site, München
- Russia (5):
  - Novartis Investigative Site, Samara, Samara Oblast
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, S-Petersburg
- Taiwan (2):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taipei

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 44 patients were randomized to receive either IV CFZ533 or IV placebo, of which 34 patients (77%) completed the study.
Pre-assignment Details: Safety analysis set, and Full analysis: 44 patients (22 treated with CFZ533 and 22 with placebo) PK analysis set : 20 patients treated with CFZ533 PD analysis set: 42 patients (20 treated with CFZ533 and 20 with placebo)
Groups:
- CFZ533: CFZ533 10 mg/kg
Period: Overall Study
Arm/Group | CFZ533 | Placebo
Started | 22 | 22
Completed | 17 | 17
Not Completed | 5 | 5
Not completed — abnormal lab value | 2 | 0
Not completed — subject / guardian decision | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CFZ533 | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (13.54) | 43.3 (13.92) | 44.0 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 10 | 6 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  caucasian | 19 | 16 | 35
  Asian (Chinese) | 3 | 5 | 8
  other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Quantitative Myastenia Gravis (QMG) Score at Week 25. Posterior Median Was Used as Measure Type.
Description: QMG score is an established validated measure of disease severity used in MG trials (Jaretzki et al 2000). The scoring system is based on quantitative testing of sentinel muscle groups by means of a 4 point scale ranging from 0 (no symptoms) to 3 (severe symptoms). The scale measures ocular, bulbar, respiratory, and limb function, grading each finding, and the total score ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits) (Sharshar et al 2000, Bedlack et al 2005).
Time Frame: week 25
Population: pharmacodynamic (PD) analysis set, participants with non-detectable AChR or MuSK autoantibodies were excluded from the PD analysis set.
Measure: Median (90% Confidence Interval); unit: score
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 18 | 18
score | -4.07 [-5.67 to -2.47] | -2.93 [-4.53 to -1.33]
Statistical Analysis 1: Comparison: CFZ533 vs Placebo; Primary analysis was performed on the PD analysis set. Changes from baseline in QMG scores at Week 25 were analyzed using a Bayesian model. The model investigated effects for treatment (CFZ533 or placebo) and baseline QMG score. A difference of 3 points on the mean change in QMG score between CFZ533 and placebo was deemed a clinical meaningful effect; Test type: Superiority; bayesian; estimate of contrast posterior median = -1.14, 90% CI 2-sided [-3.41 to 1.14]

2. Secondary Outcome: Mean Changes From Baseline in the Myasthenia Gravis Composite (MGC) Score. Posterior Median Was Used as Measure Type.
Description: The Myasthenia Gravis Composite (MGC) score is another key efficacy outcome measure, ranging from 0 to 50. It is reliable and demonstrates concurrent and longitudinal construct validity in the MG practice care setting (Burns et al 2010). The MGC scale covers 10 important functional domains most frequently involved in patients with MG. The proportion of bulbar and respiratory items reflect the clinical importance of these domains in the disease, and are appropriately weighted.
  The assessment of each of the 10 test items provides immediate insight into the status of that particular functional domain. A decrease in this score shows an improvement.
Time Frame: From baseline to week 49
Measure: Median (90% Confidence Interval); unit: score
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 18 | 18
score | -8.00 [-9.83 to -6.16] | -5.62 [-7.45 to -3.78]

3. Secondary Outcome: Proportion of Patients With Improvement or Worsening by ≥ 3 Points in the QMG Score
Description: as for outcome 1
Time Frame: at week 49
Population: PD analysis set, participants with measure
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 18 | 19
Participants
  improvement by ≥ 3 points in the QMG score | 10 | 9
  worsening by ≥ 3 points in the QMG score | 2 | 2

4. Secondary Outcome: Proportion of Patients Intolerant to Steroid Taper
Time Frame: week 49
Population: this data was not collected. No analysis could be performed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 22 | 22
Participants | NA — this data was not collected | NA — this data was not collected

5. Secondary Outcome: Number of Patients Who Discontinued Due to Inefficacy or Worsening
Time Frame: week 49
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

6. Secondary Outcome: Mean Change From Baseline in the Myasthenia Gravis-specific Activities of Daily Living Scale (MG-ADL)
Description: The MG-ADL is an 8-item survey to assess functional performance of daily activities that are sometimes impaired by MG e.g. talking, breathing, swallowing etc. (Muppidi et al 2011). The higher score on MG-ADL scale (0-24 points) indicates worse functional performance of daily activities.
Time Frame: week 25
Population: PD analysis set, participants with measure
Measure: Mean (Standard Deviation); unit: score
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 19 | 18
score | -2.6 (2.97) | -1.1 (3.23)

7. Secondary Outcome: Mean Changes From Baseline in the QMG Score at Week 49
Description: QMG (quantitative myasthenia gravis) score is an established validated measure of disease severity used in MG trials (Jaretzki et al 2000). The scoring system is based on quantitative testing of sentinel muscle groups by means of a 4 point scale ranging from 0 (no symptoms) to 3 (severe symptoms). The scale measures ocular, bulbar, respiratory, and limb function, grading each finding, and the total score ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits) (Sharshar et al 2000, Bedlack et al 2005). A decrease in the QMG score indicated an improvement. Results given as a change in the score as compared from baseline
Time Frame: week 49
Population: PD analysis set, participants with measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 18 | 19
score on a scale | -2.9 (5.16) | -2.6 (4.30)

8. Secondary Outcome: Mean Change From Baseline in the Myasthenia Gravis Quality of Life (MG QOL-15)
Description: The MG-QOL15 is a 15-item survey, completed by MG patients and it is designed to assess some aspects of quality of life (QoL) related to MG (Burns et al 2011) e.g. assesment of mood, eating, speaking, driving a car etc.. The higher score on MG-QOL15 scale (0-60 points) indicates worse QoL.
Time Frame: week 25
Population: PD analysis set, participants with measure
Measure: Mean (Standard Deviation); unit: score
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 19 | 19
score | -9.7 (11.0) | -6.7 (10.86)

9. Secondary Outcome: Free CD40 on B Cells
Description: CD40 receptor occupancy by CFZ533 in peripheral blood was assessed by flow cytometry analysis, measuring free or total CD40 receptors on whole blood B cells. Free CD40 on CD19-positive B cells, using PE-conjugated CFZ533 whose binding was prevented by bound, unconjugated CFZ533 (drug bound to CD40 on peripheral blood B cells). The more CD40 was occupied by unlabeled CFZ533, the less binding of labeled CFZ533, manifest as a lower mean fluorescence intensity (MFI) of CD40 on B cells. MFI from free CD40 on B cells was converted into Molecules of Equivalent Soluble Fluorochrome (MESF) using PE-MESF beads.
Time Frame: week 1, week 25
Population: Pharmacodynamic analysis set, participants with measure
Measure: Mean (Standard Deviation); unit: MESF
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 22 | 22
MESF
  Free CD40 on B cells week 1 predose: number analyzed (Participants) | 14 | 17
  Free CD40 on B cells week 1 predose | 34242.9 (18455.80) | 31025.9 (16138.97)
  Free CD40 on B cells week 25: number analyzed (Participants) | 8 | 12
  Free CD40 on B cells week 25 | 5259.1 (11341.57) | 24908.3 (5022.03)

10. Secondary Outcome: Total Soluble CD40 (sCD40) in Plasma
Description: PD
Time Frame: week1, week 25
Population: pharmacodynamic analysis set, participants with measure
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 22 | 22
ng/ml
  week 1: number analyzed (Participants) | 20 | 21
  week 1 | 0.1778 (0.13077) | 0.1577 (0.17243)
  week 25: number analyzed (Participants) | 18 | 19
  week 25 | 191.1278 (69.67597) | 0.1163 (0.18298)

11. Secondary Outcome: Plasma CFZ533 Concentration at Steady State Conditions (Week 17)
Time Frame: week 17
Population: pharmacokinetic set, participants treated with CFZ533 only, with measure
Measure: Mean (Standard Deviation); unit: micrograms/mL
Arm/Group | CFZ533
Number analyzed (Participants) | 18
micrograms/mL | 120 (40.5)

ADVERSE EVENTS:
Time Frame: up to week 49
Description: AE additional description
Groups:
- CFZ533 10 mg/kg IV Infusion: CFZ533 10 mg/kg IV infusion
- Placebo IV Infusion: Placebo IV infusion
Arm/Group | CFZ533 10 mg/kg IV Infusion | Placebo IV Infusion
All-Cause Mortality (participants affected / at risk) | 0/22 | 2/22
Serious Adverse Events (participants affected / at risk) | 7/22 | 4/22
Other Adverse Events (participants affected / at risk) | 20/22 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ533 10 mg/kg IV Infusion (N=22) | Placebo IV Infusion (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Influenza (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0
Brachial plexopathy (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 2 | 1
Myasthenia gravis crisis (Nervous system disorders) | 1 | 0
Radial nerve palsy (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ533 10 mg/kg IV Infusion (N=22) | Placebo IV Infusion (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 2
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Von Willebrand's disease (Congenital, familial and genetic disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Feeling cold (General disorders) | 1 | 0
Hyperthermia (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Infusion site bruising (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 2
Ear infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 1
Laryngitis viral (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 3
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 2 | 2
Rhinitis (Infections and infestations) | 1 | 0
Skin candida (Infections and infestations) | 0 | 1
Systemic infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 1 | 1
Viral pharyngitis (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Activated partial thromboplastin time shortened (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Free haemoglobin present (Investigations) | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 4 | 3
Migraine (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 2 | 1
Nerve compression (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT02565576/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT02565576/SAP_001.pdf